CLINICAL TRIAL: NCT01371292
Title: A Transformational Teaching Intervention: Adolescents in Motion (AIM) Trial
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H08-02513
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Physical Activity
Keywords: Physical activity; Transformational leadership; Physical education
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transformational teaching condition (Experimental): Teachers allocated to this condition will receive the transformational teaching intervention.
  Interventions: Behavioral: Transformational Teaching
- Standard practice control condition (Active Comparator): Teachers allocated to this condition will not receive the transformational teaching intervention. Instead they will take part in a parallel workshop offered by their respective school board (unrelated to transformational leadership training).
  Interventions: Behavioral: Standard Educational Practices

INTERVENTIONS:
Behavioral: Transformational Teaching — Physical education teachers randomly assigned to the experimental condition will (through a 1-day workshop format) be provided with the resources to implement transformational approaches in their day-to-day work. In addition, these teachers will be involved in a follow-up support program following the workshop to help them to implement transformational teaching strategies that were developed in the workshop.
  Arms: Transformational teaching condition
Behavioral: Standard Educational Practices — Physical education teachers randomly assigned to the control condition will take part in a professional development day workshop provided by their respective School Board. This will involve the same amount of contact time, and will take place on the same day as the transformational teaching workshop. It should be noted that the focus of those alternative workshops is unrelated to transformational leadership training.
  Arms: Standard practice control condition

SUMMARY:
The purpose of this Randomized Controlled Tria (RCT) is to evaluate the effects of a transformational teaching intervention in comparison to 'standard educational practices' within school-based physical education classes (within three Canadian provinces; British Columbia, Ontario and Nova Scotia) across 5 months.

DETAILED DESCRIPTION:
Physical inactivity among adolescents has been linked to a vast array of physical and mental health problems. One potential vehicle to foster adolescent involvement in physical activity relates to physical education in schools.

A potentially important framework, that has recently been applied to educational and health promotion contexts, relates to transformational leadership theory. Transformational leadership involves the demonstration of behaviors that empower and inspire others to achieve higher levels of functioning, and has been consistently found to be associated with greater motivation, self-efficacy, well-being, and performance in those being led. From an applied perspective, a growing body of evidence also suggests that transformational behaviors can be developed in leaders through short-term interventions (e.g., one-day workshops), which subsequently result in positive changes in followers' attitudinal and behavioral responses.

With this in mind, the overall goal of this Randomized Controlled Trial (RCT) is to test the efficacy of a theory-driven evidence-based transformational teaching intervention for use within school-based physical activity settings. In this 5-month trial, physical education teachers from 36 schools from three provinces across Canada (British Columbia, Ontario and Nova Scotia) will be provided with (through a one day work shop and follow-up support program) the resources they need to implement transformational teaching behaviours in their day-to-day teaching practices. The primary hypothesis for this RCT is that students taught by teachers in the intervention condition will display greater adoption and maintenance of moderate-to-vigorous physical activity (MVPA) behaviors outside of school hours in comparison to control students, after controlling for baseline levels. A process evaluation will also be conducted with teachers to evaluate the procedures embedded within the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Grade 9 (aged 14 (+/- 1 year))

Exclusion Criteria:

* Do not have basic working knowledge of English

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2160 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity (MVPA) | 5 months
  In addition to collecting self-report physical activity data through the use of questionnaires, a subsample of students (360 out of the overall sample of 2160) will be randomly selected and invited to wear a small physical activity monitor (accelerometer) on three occasions (January, March and May 2012) over the 5-month trial (for 7-days at each data point). The unit of measure that will be used to assess this outcome variable is MINUTES of moderate-to-vigorous physical activity both during leisure time hours (i.e., outside of school) and within school hours.

SECONDARY OUTCOMES:
Physical activity-related cognitions and attitudes | 5 months
  All adolescents will complete validated measures of self-efficacy (within class self-efficacy and environmental change self-efficacy), intrinsic motivation and attitudes surrounding physical education and leisure-time physical activity at each of the three time points (January, March and May 2012). Units of measure will be participants' responses on these validated scales.
Teaching efficacy | 5 months
  The physical education teachers (approximately n=72) involved in the trial will complete measures of teaching efficacy at each of the three time points (January, March and May 2012). The unit of measure will be teachers' responses on this validated scale.
Transformational teaching behaviors | 5 months
  Adolescents' perceptions of their physical education teacher's transformational behaviors will be measured at each of the three time points (January, March and May 2012). The unit of measure will be adolescents' responses on this validated scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Beauchamp, PhD, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - Acadia University, Wolfville, Nova Scotia
  - Queen's University, Kingston, Ontario
  - Nipissing University, North Bay, Ontario

REFERENCES:
- [Background] Beauchamp MR, Barling J, Li Z, Morton KL, Keith SE, Zumbo BD. Development and psychometric properties of the transformational teaching questionnaire. J Health Psychol. 2010 Nov;15(8):1123-34. doi: 10.1177/1359105310364175. Epub 2010 Jun 3. PMID 20522503
- [Background] Beauchamp MR, Morton KL. Transformational teaching and physical activity engagement among adolescents. Exerc Sport Sci Rev. 2011 Jul;39(3):133-9. doi: 10.1097/JES.0b013e31822153e7. PMID 21552132
- [Background] Morton KL, Keith SE, Beauchamp MR. Transformational teaching and physical activity: a new paradigm for adolescent health promotion? J Health Psychol. 2010 Mar;15(2):248-57. doi: 10.1177/1359105309347586. PMID 20207668
- [Background] Beauchamp MR, Barling J, Morton KL. Transformational teaching and adolescent self-determined motivation, self-efficacy, and intentions to engage in leisure time physical activity: A randomised controlled pilot Trial. DOI: 10.1111/j.1758-0854.2011.01048.x